CLINICAL TRIAL: NCT01419600
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled AZD8683 After Single Ascending Doses Administered Via Turbuhaler in Healthy Subjects
Brief Title: To Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of Inhaled AZD8683
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D1883C00006; 2011-002412-87 (EudraCT Number)
Record Dates: First submitted 2011-07-28; First posted 2011-08-18 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Phase 1; healthy volunteers; safety; tolerability; pharmacokinetics; single ascending dose study

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group 1 - 4, single ascending dose AZD 8683 (Experimental): Subjects will participate in 1 of 4 groups. In each group, 6 subjects will receive AZD8683 and 2 subjects will receive placebo.
  Interventions: Drug: AZD8683
- Group 1-4 single ascending dose Placebo (Placebo Comparator): Subjects will participate in 1 of 4 groups. In each group, 6 subjects will receive AZD8683 and 2 subjects will receive placebo.
  Interventions: Drug: Placebo to match

INTERVENTIONS:
Drug: AZD8683 — Single Dose Inhaled IMP via Turbuhaler
  Arms: Group 1 - 4, single ascending dose AZD 8683
Drug: Placebo to match — Single dose Inhaled Placebo via Turbuhaler
  Arms: Group 1-4 single ascending dose Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of increasing single doses of AZD8683 administered via inhalation

DETAILED DESCRIPTION:
A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of inhaled AZD8683 after Single Ascending Doses administered via Turbuhaler in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures Healthy male subjects aged 18
* 45 years with suitable veins for cannulation or repeated venepuncture
* Male subjects should be willing to use barrier contraception ie, condoms and spermicide, from the day of dosing until at least 3 months after dosing with the investigational product
* Have a body mass index (BMI) between 19 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive

Exclusion Criteria:

* History or presence of gastrointestinal, pulmonary, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the investigational product
* Abnormal vital signs, after 10 minutes supine rest, defined as any of the following:

  * Systolic blood pressure >140 mm Hg
  * Diastolic blood pressure >90 mm Hg
  * Heart rate <40 or >85 beats per minute Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG. This includes subjects with any of the following:
  * PR(PQ) interval prolongation >200 ms or dropped beats (single non conducted P-waves) based on screening or Prolonged QTcF >450 ms or shortened QTcF <340 ms or family history of long QT syndrome

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of AZD8683 by assessing the frequency of adverse events | Adverse events are captured from screening and captured on each clinic day and on the follow up day.
Evaluate the safety of AZD8683 by assessing a panel of laboratory safety assessments | Lab safety assessments are taken at screening, pre-dose on day 1 and then 24 hours, and 48 hours post-dose and again on follow up.
Evaluate the safety of AZD8683 by assessing dECG. | dECG is conducted pre-dose and then 15 minutes, 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 8 hours 12 hours, 24 hours and 48 hours post dose.
Evaluate the safety of AZD8683 by assessing physical examination | A physical examination is conducted at screening, day -1, day 3 and again at follow-up.
Evaluate the safety of AZD8683 by assessing vital signs (BP and pulse) | Vital signs are measured at screening, pre-dose and then 15 minutes, 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours and 48 hours post dose
Evaluate the safety of AZD8683 by assessing Spirometry | Spirometry is conducted pre-dose and at 5 minutes, 15 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours and 24 hours

SECONDARY OUTCOMES:
The maximum plasma concentration (Cmax) will be determined for AZD8683 | pre-dose and than 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours and 120 hours post dose
The time to Cmax (tmax) will be determined for AZD8683 | pre-dose and then 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours and 120 hours post dose.
The Terminal half-life (t1/2z)will be determined for the AZD8683 | pre-dose and then 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours and 120 hours post dose.
Area under the plasma concentration-time curve from zero to 24 h (AUC(0-24)) | pre-dose and than 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours post dose
Area under the plasma concentration-time curve from zero to 48 h (AUC(0-48) | 0 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours post dose
Area under the plasma concentration-time curve from zero to the time of the last measurable concentration (AUC(0-t)) | 0 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours and 120 hours post dose
Area under the plasma concentration-time curve from zero to infinity (AUC) | 0 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours and 120 hours post dose
Apparent plasma clearance (CL/F) | 0 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours and 120 hours post dose
Apparent volume of distribution during terminal phase (Vz/F) | 0 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours and 120 hours post dose
Mean residence time (MRT) | 0 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours and 120 hours post dose
Amount of drug excreted unchanged into urine in a collection interval (Ae) | 0 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours and 120 hours post dose
Fraction of dose excreted unchanged in urine (Ae/Dose) | 0 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours and 120 hours post dose
Cumulative amount of drug excreted unchanged into urine from zero to time 48 h (Ae(0-48)) | 0 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours post dose
To investigate the pharmacodynamics (PD) of inhaled single ascending doses of AZD8683 in healthy subjects including the Forced Expiratory Volume in 1 second (FEV1) | Spirometry for FEV1 is conducted pre-dose and at 5 minutes, 15 minutes, 1 hour, 2 hours and 4 hourspost dose.
To investigate the pharmacodynamics (PD) of inhaled single ascending doses of AZD8683 in healthy subjects the Forced Vital Capacity (FVC) parameter | Spirometry for FVC is conducted pre-dose and at 5 minutes, 15 minutes, 1 hour, 2 hours and 4 hourspost dose.
To investigate the pharmacodynamics (PD) of inhaled single ascending doses of AZD8683 in healthy subjects the heart rate will be measured | Heart rate is measured pre-dose and then at 15 minutes, 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours and 4 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, Study Director — AstraZeneca; Darren Wilbraham, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, London, UK, United Kingdom